CLINICAL TRIAL: NCT06934252
Title: A Phase 1a/1b Randomized, Double-Blind, Placebo-Controlled, 3-Part Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Subcutaneous Doses of TRB-061 in Healthy Participants and in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Phase 1a/1b Study of TRB-061 in Healthy Participants & Atopic Dermatitis Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TRex Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRB061-AD-101
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SAD - TRB-061 (Experimental): Single ascending subcutaneous doses of TRB-061 in healthy participants across 6 cohorts
  Interventions: Drug: TRB-061
- MAD - TRB-061 (Experimental): Multiple subcutaneous doses (Q4W for 8 weeks) in healthy participants
  Interventions: Drug: TRB-061
- MAD+ - TRB-061 (Experimental): Multiple subcutaneous doses (Q4W for 12 weeks) in patients with moderate-to-severe AD
  Interventions: Drug: TRB-061
- Placebo Comparator (Placebo Comparator): Subcutaneous placebo (matching TRB-061 in each study part
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRB-061 — Single subcutaneous injection of TRB-061 at escalating doses
  Arms: SAD - TRB-061
Drug: TRB-061 — Subcutaneous TRB-061 administered every 4 weeks for a total of 4 doses
  Arms: MAD+ - TRB-061
Drug: TRB-061 — Subcutaneous TRB-061 administered every 4 weeks for 3 doses
  Arms: MAD - TRB-061
Drug: Placebo — Single and multiple Subcutaneous doses of placebo matching TRB-061 in patients.
  Arms: Placebo Comparator

SUMMARY:
This Phase 1a/1b randomized, double-blind, placebo-controlled study evaluates the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of subcutaneously (SC) administered TRB-061 in healthy adults and patients with moderate-to-severe atopic dermatitis (AD).

Part 1 (SAD): Healthy participants receiving single doses or placebo. Part 2 (MAD): Healthy participants receiving multiple doses (3 doses over 8 weeks) of TRB-061 or placebo.

Part 3 (MAD+): Participants with moderate-to-severe AD receiving repeated doses (4 doses over 12 weeks) of TRB-061 or placebo.

DETAILED DESCRIPTION:
The study comprises three sequential parts:

Part 1 (SAD): Healthy adults will receive single-ascending doses of TRB-061 or placebo in cohorts of 8 (6 active, 2 placebo). Safety data will be reviewed before dosing the remaining participants. Follow-up lasts 12 weeks post-dosing.

Part 2 (MAD): Two cohorts of healthy adults will receive multiple doses of TRB-061 or placebo every 4 weeks (Q4W) over 8 weeks. Follow-up lasts 10 weeks post-last dose.

Part 3 (MAD+): Participants with moderate-to-severe AD will be randomized (1:1:1) to receive one of two doses of TRB-061 or placebo for 12 weeks. Responders will be followed for 36 weeks post-treatment. Non-responders will complete the study at 16 weeks. Placebo non-responders may receive 12 weeks of active treatment with a 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 to 70 years, inclusive, at the time of informed consent.
2. Body weight ≥50 kg and body mass index (BMI) between 18.5 and 35.0 kg/m², inclusive.
3. Participant is in good general health as determined by the investigator, based on medical history, physical examination, and clinical laboratory tests.
4. For healthy participants (Parts 1 and 2): no clinically significant abnormalities in laboratory results, ECGs, or physical exams at screening.
5. For participants in Part 3: diagnosis of moderate-to-severe atopic dermatitis for at least 12 months before screening.
6. Must be nonpregnant and nonlactating with negative pregnancy tests at screening and prior to dosing.
7. Must be a non-smoker or ≤5 cigarettes per week for the past 6 months.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may put the participant at risk or interfere with study results.
2. History or presence of any condition requiring systemic immunosuppressive or immunomodulatory therapy within a defined period before screening.
3. Use of any biologic agent (e.g., monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) before Day 1.
4. Participation in another investigational drug trial within 30 days or 5 half-lives of the investigational product (whichever is longer) before Day 1.
5. History of hypersensitivity or allergic reaction to any component of the study drug or placebo formulation.
6. Known active or latent tuberculosis (TB) infection or history of incomplete TB treatment.
7. Positive test at screening for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) RNA, or human immunodeficiency virus (HIV).
8. Active infection or history of serious infections within 4 weeks prior to Day 1.
9. History of malignancy (except treated and cured non-melanoma skin cancers or cervical carcinoma in situ).
10. Pregnant or breastfeeding women, or women planning to become pregnant during the study or within a specified time after the last dose.
11. Clinically significant ECG abnormalities (e.g., QTcF >470 ms) or other cardiac risk factors.
12. Abnormal laboratory values at screening
13. Use of live vaccines within 4 weeks before Day 1.
14. Use of systemic corticosteroids, immunosuppressants, or immunomodulatory drugs within protocol-defined washout periods.
15. Active COVID-19 infection or symptoms, or positive COVID-19 test at screening.
16. History of alcohol or drug abuse within the past year.
17. Use of tobacco/nicotine products beyond protocol-allowed limits.
18. Positive cotinine test at check-in.
19. Any other reason, in the opinion of the investigator or sponsor, that would make the participant unsuitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2027-06-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Screening to Day 85 (Part 1), Up to Day 127 (Part 2); up to Week 49 (Part 3)

SECONDARY OUTCOMES:
Pharmacokinetic (Maximum Observed Plasma Concentration, Cmax) | Up to Day 85 (Part 1), Up to Day 127 (Part 2); up to Week 49 (Part 3)

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No